CLINICAL TRIAL: NCT00002823
Title: A LARGE-SCALE TRIAL EVALUATING ADJUVANT CHEMOTHERAPY AFTER CURATIVE RESECTION OF NON-SMALL CELL LUNG CANCER
Brief Title: Combination Chemotherapy Compared With No Treatment Following Surgery in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065002; FRE-IALT; EU-96010
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2011-04

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage III non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cisplatin; Etoposide; Vinblastine; Vindesine; Vinorelbine; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Drug: vinblastine sulfate
Drug: vindesine
Drug: vinorelbine tartrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if combination chemotherapy given after surgery is more effective than surgery alone for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy following surgery with that of surgery alone in treating patients who have stage I, stage II, or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the impact on overall survival of adjuvant cisplatin and either a vinca alkaloid or etoposide (with or without radiotherapy) vs. no adjuvant chemotherapy in patients with completely resected stage I/II/III non-small cell lung cancer. II. Assess the frequency of treatment-related deaths and severe toxic effects. III. Describe the patterns of failure, second malignancies, and toxic effects associated with each treatment regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating institution, type of prior surgery, and pathologic stage. Each participating center will determine which combination chemotherapy regimen and which of three cisplatin doses will be given to all patients treated at that center. The treatment group receives cisplatin combined with either vindesine, vinblastine, vinorelbine, or etoposide every 3-4 weeks for 3-4 courses, depending on the dose of cisplatin. The second group receives no adjuvant chemotherapy. Treating institutions determine prior to entering the trial which patients receive adjuvant radiotherapy: none; those with node-positive disease; those with N1 disease only; those with N2 disease only; or those eligible for a randomized radiotherapy trial. For patients in the treatment group, radiotherapy begins 3-4 weeks after the last course. Patients are followed at 6 months, then annually.

PROJECTED ACCRUAL: A maximum of 3,300 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented non-small cell lung cancer Any non-small cell histology eligible Pathologic stage I/II/III disease that is completely resected with microscopically clear margins within 60 days of entry (30 days preferred)

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No clear contraindication to chemotherapy No second malignancy except: Nonmelanomatous skin cancer Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior thoracic radiotherapy Surgery: Complete resection required prior to entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 1995-02; Primary Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry L. Le Chevalier, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (123):
- United States (2):
  - Comprehensive Cancer Center at JFK Medical Center, Atlantis, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
- Getlac, Buenos Aires, Argentina
- Australia (6):
  - South Eastern Sydney Area Health Service, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Western Hospital, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- AKH Vienna, Vienna, Austria
- Belgium (5):
  - A.Z. St. Jan, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - AZ Zusters Van Barmhartigheid, Ronse
  - Sint Elizabeth Ziekenhuis, Zottegem
- Brazil (4):
  - Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro
  - Porto Alegre Hospital, Porto Alegre, Rio Grande do Sul
  - Hospital A.C. Camargo, São Paulo, São Paulo
  - University of Clementino Fraga, Rio de Janeiro
- Clinica Las Nieves, Santiago, Chile
- Colombia (2):
  - Hospital Militar Central, Bogotá
  - Instituto Nacional De Cancerologia, Bogotá
- Chest Disease Clinic, Charles University, Prague (Praha), Czechia
- National Cancer Institute of Egypt, Cairo, Egypt
- Institute for Lung Diseases, Belgrade, Federal Republic of Yugoslavia
- France (45):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Paul Papin, Angers
  - C.H. Armentieres, Armentières
  - Centre Hospital General Robert Ballanger, Aulnay-sous-Bois
  - C.H. Henri Mondor, Aurillac
  - Clinique Hauts De Seine Bagneux, Bagneux
  - C.H.G. Beauvais, Beauvais
  - Hopital Avicenne, Bobigny
  - C.M.C. Du Cedre, Bois Guillaume (Rouen)
  - Institut Bergonie, Bordeaux
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Du Meridien, Cannes
  - Hopital Fontenoy, Chartres
  - Hopital Antoine Beclere, Clamart
  - Centre Hospitalier General, Compiègne
  - Hopital Intercommunal De Creteil, Créteil
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Hopital D'Etampes, Étampes
  - C.H. De Grasse, Grasse
  - Centre Hospitalier de Lagny, Lagny
  - C.H.G. Du Havre-Hopital J. Monod, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Assistance Publique Hopitaux de Marseille Hopitaux Sud, Marseille
  - C.H. Nord Mayenne, Mayenne
  - Hopital Clinique Claude Bernard, Metz
  - Centre de Radiologie et de Traitement des Tumeurs, Meudon-la-Forêt
  - Hopital Arnaud de Villeneuve, Montpellier
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Institut Mutualiste Montsouris, Paris
  - Hospital Saint-Joseph, Paris
  - Institut Curie - Section Medicale, Paris
  - Hopital Tenon, Paris
  - C.H.G. De Pau, Pau
  - Hopital Jean Bernard, Poitiers
  - CHU De Pontchaillou, Rennes
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc
  - Centre du Rouget, Sarcelles
  - C.H. De Sens, Sens
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - C.H.G. Troyes, Troyes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Greece (8):
  - University Hospital of Heraklion, Iraklion (Heraklion), Crete
  - Evangelismos Hospital, Athens
  - Athens University-Laikon General Hospital, Athens
  - Sismanoglio Hospital, Athens
  - Sotiria Hospital Chest Diseases, Athens
  - Metaxa's Memorial Cancer Hospital, Piraeus
  - University of Patras Medical School, Rio Patras
  - George Papanicolaou General Hospital, Thessaloniki
- Israel (2):
  - Kaplan Hospital, Rehovot
  - Tel-Aviv Medical Center, Tel Aviv
- Italy (11):
  - Istituto Europeo Di Oncologia, Milan
  - Federico II University Medical School, Naples
  - Ospedale Cervello, Palermo
  - Ospedale Oncologico M. Ascoli, Palermo
  - Ospedale Civile Rimini, Rimini
  - Ospedale San Filippo Neri, Rome
  - Clinica Ars Medica, Rome
  - Istituto Di Clinica Chirurgica, Torino
  - Ospedale Molinette, Turin
  - Universita Degli Studi di Udine, Udine
  - Ospedale Di Borgo Trento, Verona
- National Kinki Central Hospital, Osaka, Japan
- Lithuanian Oncology Center, Vilnius, Lithuania
- Institut National D'Oncologie, Rabat, Morocco
- Institute of Radiotherapy and Oncology, Skopje, North Macedonia
- University of Tromso, Tromsø, Norway
- Lung Centre of the Philippines, Quezon City Diliman, Philippines
- Poland (5):
  - Bialystok Medical School, Bialystok
  - Institute of Oncology, Lodz
  - Department of Children Hematology/Oncology University of Medicine Wroclaw, Wroclaw
  - K. Dluski Hospital-Medical Academy, Wroclaw
  - Regional Hospital for Lung Disease, Zdunowo
- Hospital Santa Maria, Lisbon (Lisboa), Portugal
- University of Ljubljana, Ljubljana, Slovenia
- South Africa (3):
  - Groote Schuur Hospital, Cape Town, Cape Town
  - Sandton Oncology Centre, Johannesburg
  - Park Lane Oncology Practice, Johannesburg
- Spain (3):
  - Institut Catala d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Arnau Vilanova, Valencia
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg (Goteborg)
  - University Hospital of Linkoping, Linköping
  - Lund University Hospital, Lund
  - Karolinska Hospital, Stockholm
  - University Hospital - Uppsala, Uppsala
- Switzerland (7):
  - University Hospital, Basel
  - Ospedale San Giovanni, Bellinzona
  - Ratisches Kantons und Regionalspital, Chur
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Kantonsspital, Luzern, Luzern (Lucerne)
  - City Hospital Triemli, Zurich
  - Universitaetsspital, Zurich
- Hopital Universitaire F. Bourguiba, Monastir, Tunisia

REFERENCES:
- [Background] Reiman T, Lai R, Veillard AS, Paris E, Soria JC, Rosell R, Taron M, Graziano S, Kratzke R, Seymour L, Shepherd FA, Pignon JP, Seve P. Cross-validation study of class III beta-tubulin as a predictive marker for benefit from adjuvant chemotherapy in resected non-small-cell lung cancer: analysis of four randomized trials. Ann Oncol. 2012 Jan;23(1):86-93. doi: 10.1093/annonc/mdr033. Epub 2011 Apr 6. PMID 21471564
- [Background] Hotta K, Matsuo K, Kiura K, Ueoka H, Tanimoto M. Advances in our understanding of postoperative adjuvant chemotherapy in resectable non-small-cell lung cancer. Curr Opin Oncol. 2006 Mar;18(2):144-50. doi: 10.1097/01.cco.0000208787.91947.a2. PMID 16462183
- [Background] Pignon JP, Tribodet H, Scagliotti GV, et al.: Lung Adjuvant Cisplatin Evaluation (LACE): a pooled analysis of five randomized clinical trials including 4,584 patients. [Abstract] J Clin Oncol 24 (Suppl 18): A-7008, 2006.
- [Background] Wakelee HA, Schiller JH, Gandara DR. Current status of adjuvant chemotherapy for stage IB non-small-cell lung cancer: implications for the New Intergroup Trial. Clin Lung Cancer. 2006 Jul;8(1):18-21. doi: 10.3816/CLC.2006.n.028. PMID 16870041
- [Result] Bepler G, Olaussen KA, Vataire AL, Soria JC, Zheng Z, Dunant A, Pignon JP, Schell MJ, Fouret P, Pirker R, Filipits M, Brambilla E. ERCC1 and RRM1 in the international adjuvant lung trial by automated quantitative in situ analysis. Am J Pathol. 2011 Jan;178(1):69-78. doi: 10.1016/j.ajpath.2010.11.029. Epub 2010 Dec 23. PMID 21224045
- [Result] Arriagada R, Dunant A, Pignon JP, Bergman B, Chabowski M, Grunenwald D, Kozlowski M, Le Pechoux C, Pirker R, Pinel MI, Tarayre M, Le Chevalier T. Long-term results of the international adjuvant lung cancer trial evaluating adjuvant Cisplatin-based chemotherapy in resected lung cancer. J Clin Oncol. 2010 Jan 1;28(1):35-42. doi: 10.1200/JCO.2009.23.2272. Epub 2009 Nov 23. PMID 19933916
- [Result] Voortman J, Goto A, Mendiboure J, Sohn JJ, Schetter AJ, Saito M, Dunant A, Pham TC, Petrini I, Lee A, Khan MA, Hainaut P, Pignon JP, Brambilla E, Popper HH, Filipits M, Harris CC, Giaccone G. MicroRNA expression and clinical outcomes in patients treated with adjuvant chemotherapy after complete resection of non-small cell lung carcinoma. Cancer Res. 2010 Nov 1;70(21):8288-98. doi: 10.1158/0008-5472.CAN-10-1348. Epub 2010 Oct 26. PMID 20978195
- [Result] Filipits M, Pirker R, Dunant A, Lantuejoul S, Schmid K, Huynh A, Haddad V, Andre F, Stahel R, Pignon JP, Soria JC, Popper HH, Le Chevalier T, Brambilla E. Cell cycle regulators and outcome of adjuvant cisplatin-based chemotherapy in completely resected non-small-cell lung cancer: the International Adjuvant Lung Cancer Trial Biologic Program. J Clin Oncol. 2007 Jul 1;25(19):2735-40. doi: 10.1200/JCO.2006.08.2867. PMID 17602078
- [Result] Olaussen KA, Dunant A, Fouret P, Brambilla E, Andre F, Haddad V, Taranchon E, Filipits M, Pirker R, Popper HH, Stahel R, Sabatier L, Pignon JP, Tursz T, Le Chevalier T, Soria JC; IALT Bio Investigators. DNA repair by ERCC1 in non-small-cell lung cancer and cisplatin-based adjuvant chemotherapy. N Engl J Med. 2006 Sep 7;355(10):983-91. doi: 10.1056/NEJMoa060570. PMID 16957145
- [Result] Brambilla E, Dunant A, Filipits M, et al.: Prognostic and predictive role of alterations of the P53-bax-bcl2 pathway of apoptosis in the IALT (International Adjuvant Lung Cancer Trial). [Abstract] Lung Cancer 50 (Suppl 2): A-O-021, S10, 2005.
- [Result] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- [Result] Le Chevalier T: Results of the Randomized International Adjuvant Lung Cancer Trial (IALT): cisplatin-based chemotherapy (CT) vs no CT in 1867 patients (pts) with resected non-small cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-6, 2, 2003.